CLINICAL TRIAL: NCT00680823
Title: Is Paraspinal Intramuscular Ropivacaine Injection an Effective Treatment for Headache in a Pediatric Emergency Department?
Brief Title: Study of Intramuscular Ropivacaine Injections for Treatment of Pediatric Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Hickey (Other)
Responsible Party: Sponsor-Investigator, Robert Hickey, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO08030283
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Headache; Migraine
Keywords: Headache; Migraine; Ropivacaine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ropivacaine Injections (Experimental): Intramuscular injection of the lower cervical paraspinous muscles with 1.5 mL of 0.5% ropivacaine on each side.
  Interventions: Drug: Ropivacaine
- Normal Saline Injections (Placebo Comparator): Intramuscular injection of the lower cervical paraspinous muscles with 1.5 mL of normal saline on each side.
  Interventions: Drug: Normal saline
- Observation (No Intervention): Observation for 30 minutes.

INTERVENTIONS:
Drug: Ropivacaine — 1.5 mL IM to each side in to the lower cervical paraspinous muscles x 1.
  Arms: Ropivacaine Injections
Drug: Normal saline — 1.5 mL IM to each side in to the lower cervical paraspinous muscles x 1.
  Arms: Normal Saline Injections

SUMMARY:
Objective: To determine if lower paracervical intramuscular ropivacaine injection is an effective treatment for pediatric headache in an emergency department setting.

DETAILED DESCRIPTION:
Methods: The study will be a double-blind randomized control trial. Patients will be randomly assigned to receive either intramuscular injection of the lower cervical paraspinous muscles with 1 mL of 0.5% ropivacaine on each side, placebo injections with 1 mL normal saline on each side, or no intervention at all. If randomized to an injection, the investigator and the patient will both be blinded as to the nature of the injection.

The location of the child's pain as well as severity will be assessed immediately prior to intervention and every 10 minutes for 30 minutes. If after 30 minutes relief is insufficient for discharge to home, intravenous treatment will be instituted according to current protocol. Pain will be reassessed at the time of ultimate disposition. The scale used to assess severity will vary based on the child's age.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of headache
* Age 7-17 years

Exclusion Criteria:

* Presence of fever
* meningismus
* headache that wakes the child at night
* known organic brain disease, mass, or tumor
* history of stroke
* history of allergy to ropivacaine or other aminoacyl local anesthetics
* history of liver disease
* history of impaired cardiac function
* abnormal neurologic signs
* a focal neurologic abnormality on exam that is not a known component of the child's headache syndrome
* cognitive inability to communicate the intensity of pain.
* history of shunt or other intracranial hardware

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sieminski, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 50 | 150
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (2) | 14 (2) | 15 (2) | 14 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 38 | 114
  Male | 12 | 12 | 12 | 36
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be Pain Relief Sufficient for Discharge From the Emergency Department.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation
Number analyzed (Participants) | 50 | 50 | 50
Participants | 16 | 14 | 2

2. Secondary Outcome: Number and Percent of Patients Admitted to the Hospital for Additional Therapy in Each Treatment Arm Based Upon Treating Clinicians Decision
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation
Number analyzed (Participants) | 50 | 50 | 50
Participants | 10 | 10 | 12

3. Secondary Outcome: Re-presentation to the Emergency Department With Headache Within 72 Hours of Participating in the Study
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation
Number analyzed (Participants) | 50 | 50 | 50
Participants | 7 | 7 | 4

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Ropivacaine Injections | Normal Saline Injections | Observation
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 16/50 | 11/50 | 12/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropivacaine Injections (N=50) | Normal Saline Injections (N=50) | Observation (N=50)
pain at injection site (Musculoskeletal and connective tissue disorders) | 16 | 11 | 0
neck pain at 3 days (Musculoskeletal and connective tissue disorders) | 13 | 10 | 9
neck pain at 1 month (Musculoskeletal and connective tissue disorders) | 12 | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No